CLINICAL TRIAL: NCT02297893
Title: Improving Dexterous Skills in Parkinson's Disease: A Randomized Controlled Trial
Brief Title: Improving Dexterous Skills in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Tim Vanbellingen, Dr. phil., Luzerner Kantonsspital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Luzerner Kantonsspital
Record Dates: First submitted 2014-11-17; First posted 2014-11-21 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexterity training program (HOMEDEXT) (Experimental): This program is a a high intensity training program adapted from a previously published arm ability training program
  Interventions: Behavioral: Dexterity training program (HOMEDEXT)
- Theraband training program (Active Comparator): 7 different Theraband exercises. Total duration is 30 minutes, trained 5 times a week over a period of 4 weeks
  Interventions: Behavioral: Theraband training program

INTERVENTIONS:
Behavioral: Dexterity training program (HOMEDEXT) — The dexterity training program contains 7 exercises which focus on improving fine motor skills.
  Arms: Dexterity training program (HOMEDEXT)
Behavioral: Theraband training program — The Theraband training program contains 7 exercises which focus on improving upper limb strength
  Arms: Theraband training program

SUMMARY:
Background and aim: Patients with Parkinson's disease (PD) exhibit disturbed manual dexterity. This impairment leads to difficulties in activities of daily living (ADL) such as buttoning a T-shirt or hand-writing. The aim of the present research project is to investigate the effectiveness of a high intensity home based exercise intervention focusing on fine motor skills (HOMEDEXT), in patients with PD.

Design: A single blinded randomized controlled trial (RCT) will be performed. Randomization will be done by an independent biostatistician who will use a computerized randomization protocol. A baseline assessment and a follow-up measurement 4 weeks immediately after intervention (end of rehabilitation) will be performed. A follow-up measurement, 12 weeks later, will be done to assess long-lasting effects. Assessments will be performed by investigators who are blinded for the intervention.

Participants: One hundred and four out-patients with PD will be recruited who report specific difficulties in manual dexterity when executing ADL. Intervention: The patients will be allocated to either an intervention group (n = 52) or control group (n = 52). In the intervention group PD patients will exercise, over a period of four weeks, once/day during 30 minutes a treatment with specific exercises for dexterity. The PD patients, who will be allocated to the control group, will exercise Theraband exercises.

Outcome measures: The primary outcome measures for manual dexterity will be the Nine Hole Peg test. Secondary outcome measures will be the Coin Rotation task, a sensitive screening for dexterity. Furthermore for ADL a modified version of the subscale II of the Movement Disorders Society unified Parkinson's Disease Rating Scale (MDS-UPDRS) will be used. Parkinsonian symptoms will be assessed by the MDS-UPDRS subscale III. To assess improvements in quality of life a modified version of the Parkinson's Disease Questionnaire (PDQ-39) will be used.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurodegenerative disorder that affects both motor and non-motor basal ganglia circuitry (Stern et al., 2012). The degeneration of dopaminergic neurons in the substantia nigra leads to the clinical manifestation of the cardinal motor features of PD: bradykinesia, muscle rigidity, tremor at rest and impairment of postural reflexes (Bohlhalter & Kägi, 2011). While dopaminergic therapy improves some symptoms of PD, other symptoms, such as impaired finger dexterity, may be less responsive to pharmacological treatment (Quencer et al., 2007; Gebhardt et al., 2008). Patients with PD often report difficulties in activities of daily living (ADL), such as fastening T-shirt buttons or tying shoe laces, activities which require dexterous skills (Peto et al., 2001; Nijkrake et al., 2009). The exact mechanisms for the loss in finger dexterity are not known. Elementary motor deficits such as bradykinesia (Agostino et al., 2003), reduced strength and finger torque production (Fellows et al., 1998; de Oliveira et al., 2008) certainly play a role. However, these deficits do not fully account for the motor impairment and it has been suggested that an apraxic disorder called limb kinetic apraxia, may significantly contribute to the dexterous deficits observed in PD (Quencer et al., 2007; Gebhardt et al. 2008; Vanbellingen et al., 2011, 2012).

Only limited data exist on therapeutic interventions of dexterous problems in PD (Dixon et al., 2007; Rao, 2010). However, there is increasing evidence that allied health care, which includes physical therapy (PT), speech-language therapy and occupational therapy (OT), may complement the standard pharmacological and surgical treatments (Van der Marck et al., 2009). These therapies aim to minimize the impact of the disease process, and improve the patient's participation in ADL. Two major treatment approaches are most commonly used for PD: movement strategy training and muskuloskeletal exercises (Morris et al., 2009). By using movement strategies, patients with PD may bypass the defective basal ganglia, by engaging alternative neural circuits that are still intact (frontal and parietal cortical pathways). Examples are mental rehearsing and focusing attention (Morris et al., 2009) or using sensory cues to initiate and maintain movements (Nieuwboer et al. 2007). However, a disadvantage of this treatment approaches, particularly the recruitment of frontal cortex, is its dependence on preserved cognitive abilities. As the disease progress, many patients with PD eventually develop cognitive impairments (Aarsland et al., 2010), which could negatively influence the learning of movement strategies (Nieuwboer et al., 2009). Musculoskeletal exercises aim to improve strength, joint range of movement, muscle length and endurance (Trend et al. 2002). High intensity exercise programs have been successful and showed either short or long-term effects for balance and gait for patients with PD (Hirsch et al., 2003; Morris et al., 2009; Ebersbach et al., 2010), of which most training modes were consistent with principles promoting activity-dependent neuroplasticity (Petzinger et al. 2010). Activity-dependent neuroplasticity is defined as the modifications within the central nervous system, in response to physical activity that promotes a skill acquisition process (Adkins et al., 2006). As such intensity, specificity, difficulty; and complexity of practice appear to be important parameters for driving neuroplasticity and a potential lasting effect on both brain and behavior (Petzinger et al. 2010). In contrast to the significant short and long-term improvements which were found after high intensity training for gait and balance (Hirsch et al., 2003; Morris et al., 2009; Ebersbach et al., 2010), there is little evidence for fine motor skills in patients with PD (Gauthier et al., 1987). However, no well-designed study has been conducted, so far, which focused on these aspects of motor skills in PD.

Until date no well designed trial has been performed, in patients with PD, to investigate whether a high intensity exercise program, focusing on fine motor skills, could improve dexterous skills. As described above, patients with PD often experience impaired dexterity which leads to significant disability in several ADL, contributing to a reduced quality of life. For gait and balance disorders, high intensity training programs have been shown to be successful in patients with PD, based on training modes driving activity-dependent plasticity. However, the question remains open whether a high intensity exercise program, focusing on fine motor skills, could be effective as well in patients with PD.

The aims of the present project are to assess the outcomes of a high intensity exercise intervention, focusing on fine motor skills, in in-patients with PD. The short and long-term benefits of this training program will be compared with conventional training, which patients already receive during their hospital stay. For this purposes, a single blinded randomized controlled trial (RCT) will be performed.

Based on the literature we hypothesize that the specific home based dexterity program (HOMEDEXT) will improve fine motor skills both at short term and long-term, detected by the primary outcome measurement nine-hole peg test (Earhart et al. 2011). The improved finger and hand functions will also lead to improved ADL functioning as assessed by a modified version of the subscale II of the Movement Disorders Society unified Parkinson's Disease Rating Scale (MDS-UPDRS) (Goetz et al., 2008). Furthermore, we expect that patients with PD will report a higher quality of life (QoL), as assessed by the secondary outcome measures, a modified version of the Parkinson's Disease Questionnaire (PDQ-39) (Peto et al., 2001).

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they fulfill the criteria defined by the UK Parkinson's Disease Society Brain Bank Criteria (Hughes et al. 1992), with Hoehn and Yahr stages II to IV.

Exclusion Criteria:

* Significant medical, psychiatric co-morbidity including dementia as defined by Montreal Cognitive Assessment (MOCA) (Gill et al. 2008)
* Patients who received OT in the last 12 months to avoid carryover effects
* Inability to complete questionnaires (i.e. due to cognitive problems)
* Participation in another intervention trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Nine Hole Peg Test | 2 minutes

SECONDARY OUTCOMES:
Coin Rotation task | 4 weeks
Modified MDS-UPDRS scale II | 4 weeks
PDQ-39 | 4 weeks
Dexterity Questionnaire | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: René Müri, MD, Study Chair — University of Bern
Locations (1):
- Luzerner Kantonsspital, Lucerne, Canton of Lucerne, Switzerland

REFERENCES:
- [Background] Vanbellingen T, Kersten B, Bellion M, Temperli P, Baronti F, Muri R, Bohlhalter S. Impaired finger dexterity in Parkinson's disease is associated with praxis function. Brain Cogn. 2011 Oct;77(1):48-52. doi: 10.1016/j.bandc.2011.06.003. Epub 2011 Jul 19. PMID 21775040
- [Background] Bohlhalter S. [Update on parkinson disease]. Rev Med Suisse. 2013 Jan 30;9(371):247-8. No abstract available. German. PMID 23451586